CLINICAL TRIAL: NCT06371599
Title: Comparison of the Effect of Watching Cartoons and Playing Games as Distraction Method During Peripheral Intravenous Cannula Placement on Pain and Fear in Children Aged 6-9 Years: A Randomized Experimental Study
Brief Title: The Effect of Watching Cartoons and Playing Games as Distraction Method During Peripheral Intravenous Cannula Placement on Pain and Fear in Children Aged 6-9 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Guzide UGUCU, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MersinU*GUGUCU_003
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Procedural Pain; Fear of Pain
Keywords: pain; fear; children
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The children and their parents will be blinded to the groups. The principal researchers (R1, R2) will be blinded to the research hypotheses. The opaque envelopes are stored in a locked cabinet by the researcher who performed the randomization. Data entries will be performed using the codes A and B. Codes will be shared with the researchers after statistical analyses are conducted and the research report is written.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Playing game (Experimental): The children will be asked which game they want to play before the procedure. They will start to play the game 3 minutes before the procedure.
  Interventions: Behavioral: Playing game
- Watching cartoon (Active Comparator): The children will be asked which cartoon they want to watch before the procedure. They will start to watch the cartoon 3 minutes before the procedure.
  Interventions: Behavioral: Watching cartoon

INTERVENTIONS:
Behavioral: Playing game — Active Distraction Methods
  Arms: Playing game
Behavioral: Watching cartoon — Passive Distraction Methods
  Arms: Watching cartoon

SUMMARY:
Active and passive distraction methods are frequently used in the nursing management of procedural pain in children. There are no studies comparing the effects of watching cartoon (passive) and playing game (active) as distraction methods on pain and fear associated with peripheral intravenous cannula placement in children aged 6-9 years.

This study aimed to compare the effects of playing game (active distraction) and watching cartoon (passive distraction) techniques on pain and fear during peripheral intravenous cannula placement in children aged 6-9 years.

DETAILED DESCRIPTION:
Research Hypotheses:

H1= There is a difference in the mean WB-FACES score during the procedure between the game group (GG) and the cartoon group (CG).

H2= There is a difference in the mean CFS score during the procedure between the GG and CG groups.

Design and Settings: This parallel-group randomized trial will be conducted at the invasive procedure room of the pediatrics department of a university hospital. For this experimental research, 64 children aged 6-9 years will be assigned to two groups (Game Group=GG; n = 32 and Cartoon Group=CG; n = 32) using block randomization.

Sample Size: The trial sample was calculated based on the study findings of "Ugucu, G., Uysal, D. A., Polat, O. G., Artuvan, Z., Kulcu, D. P., Aksu, D., ... & Temel, G. O. (2022). Effects of cartoon watching and bubble-blowing during venipuncture on pain, fear, and anxiety in children aged 6-8 years: a randomized experimental study. Journal of Pediatric Nursing, 65, e107-e114.". A priori power analysis was performed based on the effect size (d = 0.885, large effect) of the difference in pain scores between the groups (during the procedure). Using G*Power 3.1.9.7, the minimum sample size was calculated as 56 children, with 28 children per group, for a two-tailed hypothesis, an effect size of d = 0.885, an allocation ratio of n1/n2=1, type I error of 0.05, and a power of 90%. Considering that there may be drop-outs during the process, the number of groups was increased by 20%. The sample size of this study was determined as 64 children (32 children in each intervention group).

Data Collection Tools: Socio-Demographic Data Collection and Procedure Follow-up Form wilkk be used. It includes "age, gender, previous experience of hospitalization, experience of procedural pain in last week, analgesic administration at least six hours before the procedure, size of peripheral IV needle, area of IV blood sample, parental presence during procedure, and baseline data of pain, anxiety and fear scores of children before procedure".

The Wong-Bakers FACES® Pain Rating Scale (WB-FACES): Developed by Wong and Baker in 1981 and revised in 1983, the instrument is used to assess physical pain in people who are communicative, responsive, and aged three years and older. The scale consists of faces ranging from "Face 0= no hurt" to "Face 10=hurts worst".

The Children's Fear Scale (CFS): The instrument assessed the pain-associated fear in children. Developed by McMurty et al. (2011), the Turkish validity-reliability study of this visual scale was conducted by Özalp-Gerçeker et al. (2018) and it is scored from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome.

iPad mini: In the both group (for game and cartoon), an iPad mini will be used that had a (7.9 inch (diagonal) LED-backlit Multi-Touch display, 2048 x 1536 resolution with a density of 326 pixels per inch (ppi) with internet access.

Interventions: The invasive procedure room in the clinic which decorated with cartoon characters and ornaments on the walls will be used. The intervention can be administered to only one child at a time in the room. In routine practice, the parental presence is supported during all invasive procedures performed on children. However, the nurses' uniforms have a print/pattern of cartoon characters in the routine practice. The room will have the same characteristics for all children and their parents in terms of environmental conditions such as light, temperature, noise, and seat. Before the procedure, children's pain, and fear will be assessed after providing developmentally appropriate information. The parents will be also informed about how to support their children. The same researchers will be performed the peripheral intravenous cannula placement (R1) and observational pain and fear assessments (R2) in all children. R1 and R2 are nurses with more than five years of experience in pediatrics and degrees in scientific fields (MScN, PhD).

Cartoon Group: In the cartoon group, the cartoons that the children liked to watch will be learned from the parents before the procedure. First, the physical comfort of the children will be ensured in the invasive procedure room. The children will be asked which cartoon they want to watch before the procedure. They will start to watch the cartoon 3 minutes before the procedure. The children will be supported by their parents in holding the tablet. The procedure and the cartoon watching intervention will be terminated simultaneously.

Game Group: In the game group, the games that the children liked to play will be learned from the parents before the procedure. First, the physical comfort of the children will be ensured in the invasive procedure room. The children will be asked which game they want to play before the procedure. They will start to play the game 3 minutes before the procedure. The children will be supported by their parents in holding the tablet. The procedure and the game playing intervention will be terminated simultaneously.

Ethical Considerations: The study was granted approval by the clinical research ethics committee and written institutional permission by the hospital. Parents will be informed about the procedure and that they could withdraw from the study at any time without explanation. Written consent of parents and verbal consent of children before the study will be obtained.

Statistical Methods: The study data will be analyzed using the statistical program.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6-9 years
* Child with need or plan for the peripheral intravenous cannula placement (antecubital fossa of arm, superficial dorsal venous of hand)

Exclusion Criteria:

* Child with a neurodegenerative disease, mental retardation, vision and hearing problems, chronic, life-threatening (sepsis, shock, respiratory / cardiac arrest) or genetic disease
* Child with use of opioids, narcotics, analgesics or sedatives in the last 24 hours before the procedure

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | during the the peripheral intravenous cannula placement
  The Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Fear by Children's Fear Scale | during the the peripheral intravenous cannula placement
  The Child Fear Scale was used.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to 4 (extreme fear). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Pain assesed by Wong-Baker FACES | at 3rd minutes after the the peripheral intravenous cannula placement
  The Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Fear by Children's Fear Scale | at 3rd minutes after the the peripheral intravenous cannula placement
  The Child Fear Scale was used.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to 4 (extreme fear). Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Guzide UGUCU, PhD, MScN, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Uysal DA, Polat OG, Ugucu G, Karakul A, Olcay AZ, Tuzun O, Yigit R. A comparison of watching cartoons versus playing games as a distraction method on pain and fear of pain during peripheral intravenous cannula placement in children aged 6-9 years: A randomized experimental study. J Pediatr Nurs. 2025 Jan-Feb;80:161-166. doi: 10.1016/j.pedn.2024.11.023. Epub 2024 Nov 30. PMID 39616818